CLINICAL TRIAL: NCT06813508
Title: Prognostic Factors for the Development of Hepatocellular Carcinoma (HCC) and Indications for Liver Transplantation in Patients With Metabolic Liver Diseases (MASLD/MASH): The BOMASH Study
Brief Title: Prognostic Factors for HCC and Liver Transplantation in Patients With MASLD/MASH
Acronym: BOMASH
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: BOMASH
Record Dates: First submitted 2025-01-10; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease; Hepatocellular Carcinoma; Metabolic Dysfunction-Associated Steatohepatitis; Liver Transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Prospective Cohort: MASLD/MASH patients prospectivelly enrolled.
- Retrospective Cohort: MASLD/MASH patients retrospectivelly enrolled.

SUMMARY:
The BOMASH study is a single-center, prospective/retrospective observational study without pharmacological interventions. It will include all patients diagnosed with Metabolic-Associated Steatotic Liver Disease (MASLD/MASH), whether newly diagnosed or previously identified at the center during follow-up or as part of routine diagnostic and therapeutic care.

The aim of the study is to identify predictive factors related to the prognosis of patients with metabolic liver disease (MASLD/MASH). Specifically, the study seeks to uncover biomarkers that can identify individuals at risk of requiring a liver transplant or developing HCC.

DETAILED DESCRIPTION:
The BOMASH study is a single-center, prospective/retrospective observational study without pharmacological interventions. It will include all patients diagnosed with Metabolic-Associated Steatotic Liver Disease and Metabolic-Associated Steatohepatitis (MASLD/MASH), whether newly diagnosed or previously identified at the center during follow-ups or as part of routine diagnostic and therapeutic care. MASLD is characterized by significant variability in terms of severity and progression rates. Although a large portion of the population is at risk, only a minority develop liver-related comorbidities. Epidemiological studies reveal that patients with MASH have a higher risk of developing liver-related complications compared to those with simple steatosis (MASLD). However, the factors driving progression to MASH and its advanced stages remain unclear, and disease staging can only be accurately determined through liver biopsy. Given the large number of individuals at risk for MASLD, liver biopsy is not a feasible screening tool for widespread use. Key challenges involve understanding the biological and environmental factors that drive variability among MASLD patients and using this knowledge to develop effective methods for risk stratification, enabling targeted treatment for individuals at the highest risk.

The identification of risk factors through the combination of non-invasive tests (serum biomarkers and non-invasive techniques) can enable risk stratification for hepatocellular carcinoma (HCC) development and identify individuals who may require liver transplantation.

A study on MASLD represents a valuable tool to enhance understanding of this nosological entity and to support basic, clinical, and epidemiological research. It also benefits individuals affected by these conditions and assists national and local authorities in planning and optimizing healthcare and social services. Systematic data collection on MASLD can be instrumental in identifying previously unrecognized risk factors that may predispose individuals to more aggressive and treatment-resistant forms of the disease.

Analyzing the collected data could highlight potential common markers among patients whose MASLD diagnosis progresses to HCC and subsequently necessitates liver transplantation. These findings would provide useful prognostic factors for patient management.

In conclusion, the opportunity to longitudinally track disease progression in a large cohort of patients with chronic metabolic liver disease could pave the way for strategies that make the management of this highly prevalent condition more sustainable for national and regional healthcare systems.

Therefore, the aim of the study is to identify predictive factors related to the prognosis of patients with metabolic liver disease (MASLD/MASH). Specifically, the study seeks to uncover biomarkers that can identify individuals at risk of requiring a liver transplant or developing HCC.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of MASLD, established according to the most recent published guidelines (EASL, EASD, EASO)
* Age ≥18 years

Inclusion Criteria for Biological Sample Collection:

* Patients requiring liver biopsy for diagnostic purposes, as indicated by the most recent published guidelines (EASL, EASD, EASO)

Exclusion Criteria:

* No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be presented to every patient with a diagnosis of MASLD/MASH, either newly diagnosed or previously diagnosed at the promoting center during follow-ups or routine diagnostic-therapeutic pathways.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2043-11-20 (Estimated); Study Completion 2044-11-20 (Estimated)

PRIMARY OUTCOMES:
Number of hepatocellular carcinoma (HCC) or liver transplantation (OLT) cases and time to onset. | From enrollment to november 2044
  The aim of the study is to identify predictive factors related to the prognosis of patients with liver disease of dysmetabolic origin: Metabolic-Associated Steatotic Liver Disease and Metabolic-Associated Steatohepatitis (MASLD/MASH). Specifically, the aim is to identify markers that can predict individuals who will later require a liver transplant or develop hepatocellular carcinoma.

SECONDARY OUTCOMES:
Incidence of HCC and liver transplantation (OLT) | From enrollment to november 2044
  Calculate the incidence of liver transplantation and the occurrence of HCC for this disease.
Response rate in patients | From enrollment to november 2044
  Objective response rate in patients with HCC or those requiring liver transplantation, measured using RECIST 1.1 criteria.
Number of cases of liver complications | From enrollment to november 2044
  Cases of liver decompensation, major adverse cardiovascular events (MACE), extrahepatic tumors, and liver transplantation, along with their time of onset.
Response to dietologic and pharmacological therapies related to glycated hemoglobin levels | From enrollment to november 2044
  Positive response to dietetic and drug therapies is measured by glycated hemoglobin levels.
Response to dieto-therapeutic and pharmacological therapies related to weight | From enrollment to november 2044
  Positive response to dietetic and pharmacological therapies is measured by weight loss.
Response to dieto-therapeutic and pharmacological therapies related to biochemical parameters | From enrollment to november 2044
  Positive response to dietetic and pharmacological therapies is measured by biochemical parameters (Aspartate amino transferase, Alanina amino transferase).
Number of HCC or liver transplantation (OLT) cases categorized by MASLD and MASH | From enrollment to november 2044

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Piscaglia, Prof, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No